CLINICAL TRIAL: NCT05881915
Title: Epinephrine Versus Phenylephrine Infusion for Prophylaxis Against Maternal Hypotension After Spinal Anesthesia for Cesarean Delivery: a Randomized Controlled Trial.
Brief Title: Epinephrine Infusion for Prophylaxis Against Maternal Hypotension After Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hassab elnaby, assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-245-2022
Record Dates: First submitted 2023-03-26; First posted 2023-05-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hypotension During Surgery
MeSH Terms: interventions — Phenylephrine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- phenylephrine (Active Comparator)
  Interventions: Drug: Phenylephrine
- epinephrine (Active Comparator)
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Phenylephrine — phenylephrine infusion at rate of 0.4 mcg/Kg/min. (10 mg /1 mL) will be diluted to reach a final concentration of 10 mcg/mL
  Arms: phenylephrine
Drug: Epinephrine — epinephrine infusion dose of 0.03 mcg/Kg/min. epinephrine (1mg/ 1mL ampoule) will be diluted to reach a final concentration of 10 mcg/ml.
  Arms: epinephrine

SUMMARY:
Subarachnoid block is the common route of anesthesia for cesarean delivery. Maternal hypotension after subarachnoid block is very common despite the vigorous methods for its prevention. Maternal hypotension is sometimes deleterious to the mother and the fetus; thus, it is highly recommended to use prophylactic vasopressors directly after the block and before the blood pressure drops. The aim of this work is to compare the maternal and neonatal effects of epinephrine and phenylephrine when used as prophylactic infusion after subarachnoid block for cesarean delivery.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitoring will be applied (electrocardiography, pulse oximetry, and a non-invasive blood pressure monitor). Two 18G-cannula will be inserted, and 10 mg metoclopramide and 50 mg ranitidine will be delivered. Co-load infusion of lactated Ringer's solution will be infused at a rate of 15 mL/Kg over 10 minutes, and 10 mg hyperbaric bupivacaine in addition to 20 mcg fentanyl will be injected in the subarachnoid space at L3-L4 or L4-L5 interspace using 25G spinal needle.

After subarachnoid block, mothers will be placed in a supine position with left-lateral tilt and will receive the vasopressor infusion according to the allocated study group:

* Phenylephrine group (n=113): will receive phenylephrine infusion at rate of 0.4 mcg/Kg/min. (10 mg /1 mL) will be diluted to reach a final concentration of 10 mcg/mL(5).
* Epinephrine group (n=113): will receive epinephrine infusion dose of 0.03 mcg/Kg/min. epinephrine (1mg/ 1mL ampoule) will be diluted to reach a final concentration of 10 mcg/ml.

The prophylactic vasopressor infusion will be maintained until 5 minutes after delivery of the fetus

Hemodynamic management in both groups will be as follow:

Post-spinal hypotension (defined as systolic blood pressure ≤80% of the baseline reading during the period from intrathecal injection to delivery of the fetus) will be managed by either ephedrine 9 mg bolus (if the heart rate was below 75 bpm) or phenylephrine 50 mg bolus (if the heart rate was above 75 bpm).

Severe post-spinal hypotension (defined as systolic blood pressure ≤60% of the baseline reading) will be managed by administration of either ephedrine 15 mg (if the heart rate was below 75 bpm) or phenylephrine 100 mg bolus (if the heart rate was above 75 bpm).

Reactive hypertension (defined as systolic blood pressure ≥120% from the baseline reading) will be managed by stoppage of the infusion till the next systolic blood pressure reading. The infusion will be then re-started at a reduced rate (50% of the initial dose) when systolic blood pressure will have decreased to be within 20% of the baseline reading.

Intraoperative bradycardia (defined as a heart rate less than 55 bpm) will be managed by stoppage of the vasopressor infusion if not associated with hypotension. The infusion will be then re-started at a reduced rate (50%) when the heart rate is more than 55 bpm. IV atropine bolus (0.5 mg) will be administered if bradycardia persisted despite stoppage of the infusion. If accompanied with hypotension, bradycardia will be managed by IV bolus of ephedrine 9 mg.

Fluid administration will be continued up to a maximum of 1.5 liters. After delivery, an oxytocin bolus (0.5 IU) will be delivered over five seconds, followed by infusion at a rate of 2.5 IU/hour.

ELIGIBILITY:
Inclusion Criteria:

* full-term singleton pregnant women, admitted for elective cesarean delivery
* aged between 18 and 40 years

Exclusion Criteria:

* Patients with uncontrolled cardiac morbidities, hypertensive disorders of pregnancy
* Peripartum bleeding
* coagulation disorders
* Baseline systolic blood pressure (SBP) < 100 mmHg

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
incidence of post spinal hypotension | from spinal anesthesia till delivery of fetus (about 45-60 mins)
  systolic blood pressure ≤80% of the baseline reading during the period from intrathecal injection to delivery of the fetus

SECONDARY OUTCOMES:
incidence post spinal reactive hypertension | from spinal anesthesia till delivery of fetus (about 45-60 mins)
  defined as systolic blood pressure ≥120% from the baseline reading
fetal outcome | at birth
  arterial blood gas

OTHER OUTCOMES:
fetal outcome | at 1 min , and at 5 min
  APGAR score (Appearance - Pulse - Grimace - Activity -Respiration ) normal 7-10
bradycardia | from spinal anesthesia till delivery of fetus (about 45-60 mins)
  heart rate less than 55 bpm

CONTACTS AND LOCATIONS:
Locations (1):
- Yasmin Ibrahim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassabelnaby YS, Hasanin AM, Shamardal M, Mostafa M, Zaki RM, Elsherbiny M, Refaat S. Epinephrine vs. phenylephrine infusion for prophylaxis against maternal hypotension after spinal anesthesia for cesarean delivery: a randomized controlled trial. J Anesth. 2024 Aug;38(4):500-507. doi: 10.1007/s00540-024-03344-2. Epub 2024 May 25. PMID 38789602